CLINICAL TRIAL: NCT02728258
Title: A Phase II Evaluation of Copanlisib (BAY 80-6946), a Selective Inhibitor of PI3KCA, in Patients With Persistent or Recurrent Endometrial Carcinoma Harboring PIK3CA Hotspot Mutations
Brief Title: Copanlisib in Treating Patients With Persistent or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GY008; NCI-2016-00325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-DT1419; NRG-GY008; NRG-GY008 (Other: NRG Oncology); NRG-GY008 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-11

CONDITIONS: Endometrial Endometrioid Adenocarcinoma; Endometrial Mixed Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Undifferentiated Carcinoma; Metastatic Endometrioid Adenocarcinoma; Recurrent Uterine Corpus Cancer
MeSH Terms: conditions — Carcinoma, Endometrioid | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (copanlisib) (Experimental): Patients receive copanlisib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Copanlisib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Copanlisib — Given IV
  Other Names: BAY 80-6946; PI3K Inhibitor BAY 80-6946
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well copanlisib works in treating patients with endometrial cancer that has not decreased or disappeared, and the cancer may still be in the body despite treatment (persistent) or has come back (recurrent). Copanlisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of copanlisib (BAY 80-6946) in patients with persistent or recurrent endometrial carcinoma harboring phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PI3KCA) hotspot mutations with the frequency of objective response.

SECONDARY OBJECTIVES:

I. To estimate 6 month progression-free survival (PFS) and median PFS. II. To estimate the distribution of the duration of overall survival (OS). III. To assess the safety profile of copanlisib in endometrial cancer patients.

TERTIARY OBJECTIVES:

I. To systematically evaluate by sequencing the site (i.e., exome) and characteristics of PIK3CA mutations in endometrial cancer patients and correlate such mutations to overall response (OR), PFS, and OS in patients treated with copanlisib.

OUTLINE:

Patients receive copanlisib intravenously (IV) over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the psychological ability and general health that permits completion of the study requirements and required follow-up
* Women of child-bearing potential (WOCBP) must agree to use adequate contraception when sexually active; patients should continue contraception for 6 months after finishing study drug
* Submission of tumor tissue is required for all patients; investigators should check with their site pathology department regarding release of biospecimens before approaching patients about participation in the trial
* Patients must have recurrent or persistent endometrial cancer (endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, mixed epithelial carcinoma or adenocarcinoma not otherwise specified [NOS]); histologic confirmation of the primary tumor is required
* All patients must have a somatic PIK3CA gene mutation (i.e., R88Q in exon 1, N345K in exon 4, C420R in exon 7, E542K, E545X [E545A, E545D, E545G, and E545K], Q546X [Q546E, Q546K, Q546L, and Q546R] in exon 9, and M1043I, H1047X [H1047L, H1047R, and H1047Y], or G1049R in exon 20) in a representative primary or metastatic tumor sample confirmed by the Roche COBAS PIK3CA Mutation Test at Q^2 Solutions
* All patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as 'non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must have recovered from effects of recent surgery, radiotherapy, or chemotherapy; at least 4 weeks must have elapsed since the patient underwent any major surgery (e.g., major: laparotomy, laparoscopy); there is no delay required for minor procedures (e.g., tumor fine-needle aspiration [FNA] or core biopsy, venous access device placement)
* Patients may have received prior radiation therapy for treatment of endometrial cancer; prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para-aortic radiation therapy, intravaginal brachytherapy and/or palliative radiation therapy; all radiation therapy must be completed at least 4 weeks prior to registration
* Patients may have received prior hormonal therapy for treatment of endometrial carcinoma; all hormonal therapy must be discontinued at least 4 weeks prior to registration
* Patients may have received prior therapy (including chemotherapy, biologic/targeted therapy and immunotherapy) for treatment of endometrial cancer; all therapy must be discontinued at least 4 weeks prior to registration; any investigational agent must be discontinued at least 30 days prior to registration
* Patients must have had at least one prior chemotherapeutic regimen for management of endometrial carcinoma; initial treatment may include chemotherapy, chemotherapy and radiation therapy, or consolidation/maintenance therapy; chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen

  * Patients are allowed to receive, but not required to receive, up to a total of 3 lines of chemotherapy
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination within 28 days prior to registration
  * Imaging of target lesion(s) within 28 days prior to registration
  * Completion of pre-study protocol specific assessments as required
* Performance status (Eastern Cooperative Oncology Group [ECOG]/Karnofsky) of 0, 1 or 2 within 28 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelets >= 75,000/mcl
* Hemoglobin (Hgb) >= 8 g/dL
* Creatinine =< 1.5 x upper limit of normal (ULN)
* Bilirubin =< 1.5 x ULN (=< 3 x ULN for patients with Gilbert syndrome)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Left ventricular ejection fraction (LVEF) >= 50%
* Fasting cholesterol less than or equal to 300 mg/dl; fasting triglycerides less than or equal to 300 mg/dl
* Prothrombin time (PT) such that international normalized ratio (INR) is less than or equal to 1.5 x ULN (or an in range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) less than or equal to 1.5 times the upper limit of normal
* The patient must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information
* Diabetic patients (type I or II diabetes mellitus) must have baseline hemoglobin (Hb)A1c levels NOT higher than 8.5% at study entry
* Patients with hypertension on medical management must have systolic blood pressure < 150 mmHG or diastolic pressure < 90 mmHG at study entry
* Note: ULN is institutional or laboratory upper limit of normal
* Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test within 28 days of registration; the patient and her sexual partner(s) must agree to use adequate contraception when sexually active for the duration of the study and for 6 months after finishing study drug; a woman is considered of childbearing potential following menarche and until becoming post-menopausal unless permanently sterile; permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy; a postmenopausal state is defined as no menses for 12 months without an alternative medical cause; a high follicle stimulating hormone (FSH) level in the postmenopausal range maybe used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy

Exclusion Criteria:

* Patients who have had prior therapy with any phosphatidylinositol 3 kinase (PI3K)/v-akt murine thymoma viral oncogene homolog 1 (AKT)/mammalian target of rapamycin (mTor) pathway inhibitor
* Patients who have the following histologies: mucinous, squamous, sarcomas, carcinosarcomas, clear cell
* Congestive heart failure > New York Heart Association (NYHA) class II
* Myocardial infarction or unstable angina less than 6 months before registration
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before registration
* Non-healing wound, ulcer or bone fracture
* Active, clinically serious infections > Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* History of, or current autoimmune disease
* Human immunodeficiency virus (HIV) infection
* Hepatitis B (HBV) or hepatitis C (HCV); all patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus laboratorial panel; patients with active HBV or hepatitis C infection are not eligible for enrollment; patients with serologic markers of HBV immunization due to known vaccination (hepatitis B surface antigen [HBsAg] negative, anti-hepatitis B core [HBc] negative and anti-hepatitis B surface [HBs] positive) will be eligible
* Previous or concurrent history of malignancies within 5 years prior to study treatment except for curatively treated:

  * Cervical carcinoma in situ
  * Non-melanoma skin cancer
  * Superficial bladder cancer (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria])
* Patients with seizure disorder requiring medication
* Patients with evidence or history of bleeding diathesis; any hemorrhage or bleeding event >= CTCAE grade 3 within 4 weeks prior to registration
* Proteinuria of CTCAE grade 3 or higher (estimated by urine protein: creatinine ratio >= 3.5 on a random urine sample); patients who recently (i.e., at least 30 days prior to registration) discontinued an anti-angiogenic therapy which caused proteinuria (ie, grade 2 (> 2 to > 3 g of protein or 1-3.5 g/24 hours [h]) or grade 3 proteinuria (> 4 of protein or > 3.5 g/24 h) are not eligible for enrollment until proteinuria improves to < 2 g of protein per 24 h
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
* Concurrent diagnosis of pheochromocytoma
* Unresolved toxicity higher than CTCAE grade 1 attributed to any prior therapy/procedure, excluding alopecia
* Known hypersensitivity to any of the test drugs, test drug classes, or excipients in the formulation
* Strong CYP3A4 inhibitors and inducers; concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and inducers of CYP3A4 (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) are not permitted within two weeks prior to start of study treatment and for the duration of treatment with copanlisib
* Grapefruit and grapefruit juice (CYP3A4 inhibitor), Seville oranges and star fruit consumption is not permitted during the study
* Anti-arrhythmic therapy other than beta blockers or digoxin
* Systemic continuous corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not allowed; patients may be using topical or inhaled corticosteroids
* Concomitant therapy with any anticancer agents, immunosuppressive agents, other investigational anticancer therapies
* Concomitant radiotherapy
* Women who are breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D Santin, Principal Investigator — NRG Oncology
Locations (43):
- United States (43):
  - Yale University, New Haven, Connecticut
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Northside Hospital, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Baystate Medical Center, Springfield, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated 9/16/2016 and the last patient was enrolled in May 2017. The study was officially closed to accrual on 8/7/2017 after the first stage of accrual was completed and all screened patients were either enrolled or refused. The study did not continue on to the second stage of accrual.
Pre-assignment Details: Tumor samples were screened for somatic "hotspot" PIK3CA gene mutations prior to enrollment.
Groups:
- Copanlisib: IV copanlisib (60 mg weekly, day 1, 8 and 15 of 28-day cycle)
Period: Overall Study
Arm/Group | Copanlisib
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All eligible and evaluable participants
Arm/Group | Copanlisib
Number analyzed (Participants) | 11
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 3
  60-69 years | 4
  70-79 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Objective Response Defined by RECIST 1.1 Criteria
Description: Confirmed complete and partial tumor response by RECIST 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: approximate study duration 1 year 9 months
Population: Eligible and treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Copanlisib
Number analyzed (Participants) | 11
percentage of participants | 0.0 [0 to 28.5]

2. Secondary Outcome: Percentage of Participants Alive and Progression-free at 6 Months
Description: Percentage of participants who are progression free at 6 months. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 6 months from enrollment
Population: Eligible and treated patients
Measure: Number; unit: percentage of participants
Arm/Group | Copanlisib
Number analyzed (Participants) | 11
percentage of participants | 27

3. Secondary Outcome: Median Progression-Free Survival Using RECIST 1.1 Criteria
Description: The median progression-free survival time
Time Frame: Up to 2 years from enrollment
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Copanlisib
Number analyzed (Participants) | 11
Months | 2.8 [1.6 to 8.9]

4. Secondary Outcome: Median Overall Survival
Description: Median time of overall survival
Time Frame: up to 2 years from enrollment
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Copanlisib
Number analyzed (Participants) | 11
Months | 15.2 [4.7 to 21]

5. Secondary Outcome: The Frequency and Severity of CTCAE v4 Graded Adverse Events
Description: Maximum grade of physician assessed adverse events reported during treatment
Time Frame: approximately 1 year 9 months
Population: Eligible and treated patients
Measure: Number; unit: participants
Arm/Group | Copanlisib
Number analyzed (Participants) | 11
participants
  Grade 1 | 1
  Grade 2 | 1
  Grade 3 | 7
  Grade 4 | 2
  Grade 5 | 0

6. Other Pre Specified Outcome: Mutation Subtypes and Clinical Outcomes
Description: Associations between mutation subtypes and clinical outcomes will be explored using standard statistical methods for categorical and time to event data.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed throughout the treatment period and up to 4 weeks after discontinuation of treatment
Arm/Group | Treatment (Copanlisib)
All-Cause Mortality (participants affected / at risk) | 7/11
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Copanlisib) (N=11)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cellulitis (other) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Copanlisib) (N=11)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (4)
Rectal Pain (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4)
Oral Dysesthesia (Gastrointestinal disorders) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Chills (General disorders) | 1 (1)
Edema Limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Fever (General disorders) | 1 (1)
Infusion Related Reaction (General disorders) | 2 (2)
Localized Edema (General disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin Infection (Infections and infestations) | 2 (2)
Cholesterol High (Investigations) | 1 (1)
Creatinine Increased (Investigations) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 1 (1)
Neutrophil Count Decreased (Investigations) | 3 (3)
White Blood Cell Decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Bladder Spasm (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Urinary Urgency (Renal and urinary disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
The study did not continue on to the second stage of accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT02728258/Prot_SAP_000.pdf